CLINICAL TRIAL: NCT00398645
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of GW685698X 200 mcg Twice Daily, GW685698X 200 mcg and 400 mcg Once Daily in the Morning, and GW685698X 200 mcg and 400 mcg Once Daily in the Evening Compared With Placebo for 8 Weeks in Adolescent and Adult Subjects (12 Years of Age and Older) With Persistent Asthma
Brief Title: A Randomized Study To Evaluate The Efficacy And Safety Of An Investigational Drug In Adolescent And Adult Subjects With Persistent Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FFA106783
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Asthma
Keywords: GW685698X; Adults; Pharmacokinetics; Pharmacogenetics; Asthma; Adolescents
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: GW685698X 200mcg,GW685698X 200mcg and 400mcg

INTERVENTIONS:
Drug: GW685698X 200mcg,GW685698X 200mcg and 400mcg
  Other Names: GW685698X 200mcg; GW685698X 200mcg and 400mcg

SUMMARY:
This study is designed to determine if the investigational drug is effective and safe in individuals with asthma.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of GW685698X 200mcg Twice Daily, GW685698X 200mcg and 400mcg Once Daily in the Morning, and GW685698X 200mcg and 400mcg Once Daily in the Evening Compared with Placebo for 8 Weeks in Adolescent and Adult Subjects (12 Years of Age and Older) with Persistent Asthma.

ELIGIBILITY:
Inclusion criteria:

* Type of Subject: Outpatient
* Age: 12 years of age or older at Visit 1 (or ³18 years of age or older if local regulations or the regulatory status of study medication permit enrollment of adults only).
* Gender: Male or eligible female - Females are eligible to participate only if they are currently non-pregnant and non-lactating. To be eligible for entry into the study, females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control, as defined by the following: Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject, Implants of levonorgestrel, Injectable progestogen, Oral contraceptive (either combined estrogen/progestin or progestin only), Any intrauterine device (IUD) with a documented failure rate of less than 1% per year, Double-barrier method - spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a spermicide and female diaphragm), The contraceptive transdermal patch, Ortho Evra (if the subject is less than 198 pounds), Female subjects should not be enrolled if they plan to become pregnant during the time of study participation. A urine pregnancy test is required for all subjects at all visits, Female subjects should not be enrolled if they plan to become pregnant during the time of study participation. A urine pregnancy test is required for all subjects at all visits, Female subjects should not be enrolled if they plan to become pregnant during the time of study participation. A urine pregnancy test is required for all subjects at all visits, Females of childbearing potential who are not sexually active must commit to complete abstinence from intercourse throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of six days),
* Asthma Diagnosis: Asthma as defined by the National Institutes of Health [National Institutes of Health, 2002; GINA, 2005].
* Severity of Disease: A best AM FEV1 of 50% to 80% of the predicted value during Visit 1 based on the "Standardization of Lung Function Tests" [European Respiratory Society, 1993] standards for 18 years and older or Polgar [Polgar, 1971] standards for 12 to 17 years and race adjusted for African-Americans [American Thoracic Society, 1991].
* Reversibility of Disease: Demonstrated ³12% and 200mL reversibility of FEV1 within 30 minutes following 200 to 400mcg of albuterol/salbutamol inhalation aerosol (or one nebulized albuterol/salbutamol treatment) at Visit 1. If a subject fails to demonstrate an increase in FEV1 of ³12% and 200mL, the subject is not eligible for the study and will not be allowed to re-screen.
* Concurrent Anti-Asthma Therapy: Subjects must be using an inhaled corticosteroid for at least 3 months prior to Visit 1 and be maintained on a stable dose for four weeks prior to Visit 1 at one of the following doses: Anti-Asthma Therapy Maximum Daily Dose (mcg/day) Fluticasone propionate MDI CFC/HFA ≤220mcg1/≥250mcg2 Fluticasone propionate DPI 200mcg Beclomethasone dipropionate 420mcg1/500mcg2 Beclomethasone dipropionate HFA 160mcg1/200mcg2 Budesonide DPI 400mcg Flunisolide 1000mcg Triamcinolone acetonide 1000mcg Mometasone furoate 200mcg Ciclesonide 160mcg1/200mcg2

  1. Ex-actuator dose: dose delivered to the lungs
  2. Ex-valve dose: dose expressed from the valve
* Short-Acting Beta2-Agonist: All subjects must be able to replace short-acting beta2-agonists with albuterol/salbutamol inhalation aerosol at Visit 1 for use as-needed for the duration of the study. Subjects must be able to withhold all inhaled short-acting beta-sympathomimetic bronchodilators for at least 6 hours prior to study visits.Note: Nebulized albuterol/salbutamol will not be allowed during the study with the exception of its use during reversibility testing at Visit 1. The use of albuterol/salbutamol through the DISKUS/ACCUHALER device will not be allowed during the study.
* Informed Consent: All subjects must be able and willing to give written informed consent to take part in the study.
* Compliance: Subjects must be able to comply with all the study requirements.

Exclusion criteria:

* History of Life-Threatening Asthma: History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures.
* Anti-Asthma Medications: Asthma medications listed below must not have been used prior to Visit 1 for the required interval listed below, and not taken during the study: Within 24 hours of Visit 1: Oral short-acting beta2-agonists: Within 2 weeks of Visit 1:Combination therapy containing inhaled beta2-agonists and ICS for asthma (e.g., fluticasone propionate/salmeterol combination, budesonide/formoterol combination);Slow-release bronchodilators (e.g., aminophylline, theophylline);Anticholinergics; Long-acting beta2-agonists (e.g., salmeterol); Ketotifen; Nedocromil sodium; Sodium cromoglycate; Oral long-acting beta2-agonists. Within 4 weeks of Visit 1: Anti-leukotrienes including suppressors of leukotriene production and antagonists. Within 12 weeks of Visit 1: Systemic, oral, parenteral, or depot corticosteroids; Anti-IgE (e.g., omalizumab).
* Other Medications: The medications listed below must not have been used prior to Visit 1 for the required interval indicated below, and not taken during the study: Within 4 weeks of Visit 1: Known potent inhibitors of CYP3A4 (e.g., ritonavir, ketoconazole)
* Respiratory Infection: History of a respiratory tract infection within 4 weeks of Visit 1. In addition, the subject must be excluded, if such infection occurs between Visits 1 and 2.
* Asthma Exacerbation: History of a an asthma exacerbation within 4 weeks of Visit 1, any asthma exacerbation requiring oral corticosteroids within 3 months of Visit 1, or any hospitalization due to asthma exacerbation within 6 months of Visit 1.
* Investigational Medications: A subject must not have used any investigational drug within 30 days prior to Visit 1 or within ten half-lives (t1/2) of the prior investigational study (which ever is longer of the two) or concurrently during the study.
* Concurrent Diseases/Abnormalities: Historical or current evidence of clinically significant uncontrolled disease including, but not limited to: cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, or pulmonary disease (including, but not confined to chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, bronchopulmonary dysplasia, and chronic obstructive pulmonary disease). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Oropharyngeal Examination: A subject will not be eligible for the run-in if he/she has evidence of oropharyngeal candidiasis at Visit 1.
* Drug Allergy: Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy.
* Milk Protein Allergy: History of severe milk protein allergy.
* Immunosuppressive Medications: A subject must not be using, or require use of, immunosuppressive medications during the study.

Note: Immunotherapy for the treatment of allergies is allowed during the study provided that it was initiated prior to Visit 1 and the subject is maintained on a stable daily dose throughout the study period.

* Attendance: A subject will not be eligible if he/she or his/her parent or legal guardian has any infirmity, disability, or geographical location which seems likely (in the opinion of the Investigator) to impair compliance with any aspect of this study protocol or scheduled visits to the study center and compliance with study medication or procedures (e.g., completion of daily diary). Neurological or psychiatric disease or history of drug or alcohol abuse which would interfere with the subject's proper completion of the protocol requirements excludes study participation.
* Tobacco Use: A subject may not have used tobacco products within the past one year (i.e., cigarettes, cigars, or pipe tobacco) and must not have historical use of >10 pack years (e.g., 20 cigarettes/day for 10 years).
* Affiliation with Investigator's Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2006-11-15; Primary Completion 2007-08-01 (Actual); Study Completion 2007-08-30 (Actual)

PRIMARY OUTCOMES:
The primary efficacy measure will be mean change from baseline at Week 8 (last assessment on treatment using last observation carried forward) in tough (AM or PM pre-dose and pre-rescue bronchodilator) forced expiratory volume in one second (FEV1)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (70):
- United States (16):
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Greenfield, Wisconsin
- Australia (7):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Concord, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Toorak Gardens, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Bulgaria (4):
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
  - GSK Investigational Site, Veliko Tarnovo
- Canada (3):
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Woodstock, Ontario
- Chile (3):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Croatia (2):
  - GSK Investigational Site, Split
  - GSK Investigational Site, Zagreb
- Germany (3):
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Berlin
- Israel (4):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Rehovot
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México
- New Zealand (2):
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Wellington
- Peru (2):
  - GSK Investigational Site, San Isidro, Lima region
  - GSK Investigational Site, Lima
- Philippines (3):
  - GSK Investigational Site, Cebu
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Russia (7):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Yekaterinburg
- South Africa (5):
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, eManzimtoti
  - GSK Investigational Site, Newtown
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
- Ukraine (4):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Vinnitsa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Woodcock A, Bateman ED, Busse WW, Lotvall J, Snowise NG, Forth R, Jacques L, Haumann B, Bleecker ER. Efficacy in asthma of once-daily treatment with fluticasone furoate: a randomized, placebo-controlled trial. Respir Res. 2011 Oct 6;12(1):132. doi: 10.1186/1465-9921-12-132. PMID 21977941
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: FFA106783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFA106783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFA106783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFA106783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFA106783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFA106783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFA106783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register